CLINICAL TRIAL: NCT06568328
Title: A Study to Evaluate the Safety, Tolerability, Efficacy, Pharmacokinetics and Pharmacodynamics of CNK-UT Cells to Treat the Patients With Steroid-refractory/Resistant or Steroid-dependent GVHD
Brief Title: Chimeric Natural Killer Receptor-Universal T Cells for Refractory GVHD
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Ting YANG, Prof., Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNK-UT-IIT202303
Record Dates: First submitted 2024-08-03; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Graft vs Host Disease
Keywords: Chimeric natural killer receptor universal T-cells; steroid-refractory/resistant or steroid-dependent GVHD
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CNK-UT cells therapy (Experimental): 1. Dose Escalation：Single-dose intravenous injection of CNK-UT cells (1~10×10^7 CNK+ cells/kg).
  2. Dose Expansion：Multiple-dose intravenous injection of CNK-UT cells according to the results of dose escalation.
  Interventions: Biological: Chimeric Natural Killer Receptor Universal T-cells (CNK-UT)

INTERVENTIONS:
Biological: Chimeric Natural Killer Receptor Universal T-cells (CNK-UT) — OUTLINE: This is a dose-escalation study of CNK-UT cells followed by a dose-expansion study.
  1. Dose Escalation (Single Ascending Dose Study, SAD): During SAD study stage, the participants will be intravenous infused with CNK-UT cells (1~10×10^7 CNK+ cells/kg)with a"3 +3" design to determine the maximum tolerated dose. During single ascending dose (SAD) study stage, the participants will receive a single dose of CNK-UT cells before the DLT observation period (21 days). If the participants do not experience DLT, they will be able to enter a multiple ascending dose (MAD) study stage.
  2. Dose Expansion (multiple ascending dose study, MAD): During MAD study stage, the participants will receive multiple doses of CNK-UT cells. The dosage and frequency of drug administration in the dose expansion stage can be adjusted and determined according to the SAD study.

SUMMARY:
This is a single arm, open-label, multi-center, pilot studies (Investigator Initiated Trial, IIT) to evaluate the safety, tolerability, efficacy, pharmacokinetics and pharmacodynamics of universal T-cells engineered with chimeric natural killer receptor (CNK-UT) to treat the patients with steroid-refractory/resistant or steroid-dependent GVHD.

DETAILED DESCRIPTION:
This is a single arm, open-label, phase I, dose escalation/dose expansion study to assess the safety and tolerability of CNK-UT cells therapy, and to obtain the efficacy, pharmacokinetics and pharmacodynamics result in participants who have been diagnosed with steroid-refractory/resistant or steroid-dependent GVHD.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 1~70 years, male or female;
2. Participants diagnosed with grade II~IV steroid-refractory/resistant or steroid-dependent GVHD after allogeneic hematopoietic stem cell transplantation who have failed treatment with ruxolitinib or at least one other second-line medication, or who are intolerant to these medications.
3. ECOG physical status score 0~3;
4. Estimated life expectancy > 12 weeks;
5. Female participants of childbearing age must undergo a serum or urine pregnancy test before enrollment, and the results must be negative, and agree to take acceptable measures to minimize the possibility of pregnancy during the trial; For female participants of childbearing age or male participants whose sexual partners are women of childbearing age, effective contraceptive measures should be taken during the study and for at least 6 months following the last dose of the study cells infusion.
6. Participants voluntarily participate in clinical trial; Understand and know this study, sign an informed consent form, and be willing to follow all experimental procedures.

Exclusion Criteria:

1. Suffering from malignant tumors or diagnosed within 5 years before enrollment, excluding radical skin basal cell carcinoma, skin squamous cell carcinoma, thyroid cancer, breast cancer (ductal carcinoma in situ) and / or radical resection of carcinoma in situ.
2. Participants with a history of organ transplantation;
3. Participants who have previously undergone more than one allogeneic hematopoietic stem cell transplantation.
4. Uncontrolled hypertension as determined by principal investigator, a history of hypertensive crisis or hypertensive encephalopathy; symptomatic congestive heart failure (New York Heart Association classification III-IV); symptomatic or poorly controlled arrhythmias; a history of congenital long QT syndrome or a corrected QT interval (QTc) > 500 ms at screening (calculated using the Fridericia method)..
5. Systemic diseases deemed unstable by principal investigator include, but are not limited to, severe pulmonary, hepatic, renal, or metabolic disorders that require pharmacological intervention (excluding complications related to allogeneic hematopoietic stem cell transplantation).
6. Active pulmonary tuberculosis (TB), who is receiving anti-tuberculosis treatment or has received anti-tuberculosis treatment within 1 year before enrollment; human immunodeficiency virus (HIV) infection, known syphilis infection.
7. Severe infections that are active or poorly controlled clinically.
8. Participants who have received treatment from other clinical trials within 12 weeks prior to the initiation of the study.
9. Participants who have previously used any gene therapy products prior to the initiation of the study.
10. Allergic to components of CNK-UT injection.
11. Participants suffer from known mental or substance abuse disorders, which may interfere with their ability to comply with research requirements.
12. Women who are pregnant or breastfeeding, as well as male or female participants who have planned for birth within 1 year after receiving medication.
13. Uncontrolled/uncorrectable metabolic disorders or other non-malignant organ diseases or systemic diseases or secondary reactions to cancer, which can lead to higher medical risk and/or uncertainty in survival assessments.
14. Other situations that the participant is identified by the investigator as unsuitable to participate in the study.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related adverse events (AEs) | up to 1 year
  Incidence of Treatment Related AEs, AEs of special interest and serious adverse events (SAEs) assessed by NCI-CTCAE v5.0 criteria
Identification of Maximum Tolerated Dose (MTD) & incidence of Dose-limiting Toxicities (DLTs) | up to 21 days since first infusion of CNK-UT cells
  Incidence of dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 6 months
  Overall response is defined as either a complete or partial response (CR+PR), the response should be confirmed no less than 4 weeks after the first evaluation.
Best Overall Response (BOR) | 6 months
  The best efficacy recorded from the beginning of treatment to the progression or recurrence of the disease.
Duration of Response (DOR) | 6 months
  The period from the first evaluation of CR or PR to the first evaluation of PD or death of any cause.
Progression-free Survival (PFS) | 6 months
  The period from the day when the participant receives the cell therapy to the first recorded disease progression (whether treated or not) or death of any cause, which occurs first.
Overall survival (OS) | 6 months
  The period from the first infusion to any cause of death.
Pharmacokinetics (PK) (Cmax) | up to 48 weeks
  The Peak Plasma concentration (Cmax) of amplified CNK-UT DNA in peripheral blood after infusion.
Pharmacokinetics (PK) (Tmax) | up to 48 weeks
  The time to reach the maximum concentration (Tmax)
Pharmacokinetics (PK) | up to 48 weeks
  The Area under the plasma concentration versus time curve (AUC) of amplified CNK-UT DNA in peripheral blood after infusion.
Levels of peripheral blood lymphocyte subsets | up to 48 weeks
  Percentage of CD45+CD3+TCR+T cell、CD3+CD8+ CD25+ CD69+T cell、CD3+CD4+CD25+ CD69+ T cell and Treg（CD4+CD25+FoxP3+）cell in peripheral blood detected by FCM after infusion.

OTHER OUTCOMES:
Biomarkers | Enrollment and evaluated as complete remission (CR), or if necessary，up to 48 weeks
  ST2、REG3α and Elafin will be analyzed
HLA typing | Enrollment.
  Evaluate the impact of HLA typing matching between donors and participants on the survival time and efficacy of CNK-UT in vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Ting YANG, Prof., Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China